CLINICAL TRIAL: NCT07253142
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Combination With Serplulimab (Humanized Anti-PD-1 Monoclonal Antibody Injection) in Advanced Stage Lung Cancer
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Combination With Serplulimab in Subjects With Advanced Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-NSCLC202
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX43 dose 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first).
  Interventions: Drug: HLX43 dose 1
- HLX43 dose 2 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 2

INTERVENTIONS:
Drug: HLX43 dose 1 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Serplulimab
  Arms: HLX43 dose 1
Drug: HLX43 dose 2 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Serplulimab
  Arms: HLX43 dose 2

SUMMARY:
The study is to explore the the reasonable dosage and to evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in combination with Serplulimab (anti-PD-1 humanized monoclonal antibody injection) in patients with advanced lung cancer.

DETAILED DESCRIPTION:
This study is a randomized, open-label phase II clinical study to explore the the reasonable dosage and to evaluate the efficacy, safety and tolerability of HLX43 in combination with serplulimab in patients with advanced lung cancer who have received immunotherapy and platinum-contained chemotherapy, including actionable gene alteration (AGA) negative non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC). In this study, eligible subjects will be randomized at 1:1 ratio, and the patients will be administered with HLX43 at one of the two dose levels plus serplulimab at a fixed dosage via intravenous infusion every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily to participate in the trial, and be able to complete the study as required by the protocol;
* 2. Age ≥18 years and ≤75 years;
* 3. Histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC unsuitable for radical treatment without actionable gene alteration (AGA); or Histologically or cytologically confirmed SCLC unsuitable for radical treatment, with evidence of disease progression or recurrence;
* 4. Subjects must meet the following prior treatment requirements:

  1. Have received platinum-based chemotherapy combined with anti-PD-1/L1 monoclonal or bispecific antibodies as prior first-line treatment; have received no more than second-line treatment; or
  2. Have received platinum-based chemotherapy and anti-PD-1/L1 monoclonal or bispecific antibodies (in any sequence) as sequential treatment; have received no more than third-line treatment;
* 5. Within 4 weeks prior to randomization, have at least one measurable lesion according to RECIST 1.1 efficacy evaluation criteria;
* 6. Subjects agree to provide archived tumor tissue samples (from the most recent surgery or biopsy, preferably within 2 years) that meet testing requirements or agree to undergo a biopsy to collect tumor tissue for PD-L1 expression testing;
* 7. Before the first administration of the investigational drug, there must be at least a 3-week interval or 5 half-lives of the drug (whichever is shorter) from prior major surgical procedures, device therapy, local radiotherapy (excluding palliative radiotherapy for bone lesions), cytotoxic chemotherapy, immunotherapy, or biological therapy. There must be at least a 2-week interval from prior hormone therapy or small molecule targeted therapy, and at least a 1-week interval from traditional Chinese medicine with anti-tumor indications or minor surgical procedures. Adverse events caused by prior treatment must have recovered to CTCAE v5.0 ≤ grade 1 (excluding grade 2 peripheral neurotoxicity and alopecia);
* 8. ECOG performance status score of 0-1 within one week prior to randomization;
* 9. Expected survival time of more than 3 months;
* 10. Laboratory tests within one week prior to randomization confirm adequate organ function (within 14 days before the first administration, without receiving treatments such as transfusion, granulocyte colony-stimulating factor, thrombopoietin, or erythropoietin);
* 11. Male and female subjects with reproductive potential must agree to use at least one highly effective contraceptive method during the trial and for at least 6 months after the last administration of the investigational drug. Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* 1. Mixed SCLC, mixed NSCLC, or sarcomatoid carcinoma components confirmed by tumor histology or cytology;
* 2. Imaging suggests tumor invasion of major blood vessels or important organs, or the presence of a risk of esophago-tracheal fistula or esophagopleural fistula;
* 3. Previously received any drug therapy targeting topoisomerase I, including chemotherapy or ADC drugs;
* 4. Received radical radiotherapy within 3 months prior to the first dose;
* 5. History of any second malignancy within 2 years prior to randomization, except for early-stage malignancies treated with radical therapy (carcinoma in situ or stage I tumors), such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ of the breast, or papillary thyroid carcinoma;
* 6. History of adverse events leading to permanent discontinuation of immunotherapy, or a history of ≥ grade 2 immune-related pneumonitis or immune-related myocarditis;
* 7. Presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* 8. Presence of spinal cord compression or clinically active central nervous system metastases (referring to untreated or symptomatic metastases, or metastases requiring corticosteroids or anticonvulsants to control related symptoms), or meningitis carcinomatosa. Subjects who have previously received treatment for brain metastases (e.g., whole-brain radiotherapy or stereotactic brain radiotherapy) may participate in the study, provided they have been clinically stable for at least 4 weeks with no imaging evidence of brain metastasis progression;
* 9. History or current presence of clinically severe lung impairment caused by pulmonary diseases, including but not limited to any underlying pulmonary disease (e.g., pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive pulmonary disease, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, pleural effusion, etc., within 3 months prior to the first dose) or any autoimmune, connective tissue, or inflammatory diseases potentially involving the lungs (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or subjects who have undergone pneumonectomy, which may interfere with the detection and management of suspected drug-related pulmonary toxicity; subjects with radiation pneumonitis within 6 months;
* 10. Subjects with poorly controlled cardiovascular or cerebrovascular clinical symptoms or diseases;
* 11. Presence of active systemic infectious diseases requiring intravenous antibiotic therapy within 2 weeks prior to randomization;
* 12. Use of moderate or strong CYP2D6 or CYP3A inhibitors or inducers within 2 weeks prior to randomization;
* 13. Patients who received systemic corticosteroids (prednisone >10mg/day or equivalent doses of similar drugs) or other immunosuppressive therapy within 2 weeks prior to randomization;
* 14. Presence of known active or suspected autoimmune diseases. However, patients with autoimmune-related hypothyroidism receiving thyroid hormone replacement therapy are allowed to participate in the study; patients with controlled type 1 diabetes receiving insulin therapy are allowed to participate in the study;
* 15. Received live or attenuated live vaccines within 4 weeks prior to randomization;
* 16. Known history of allergic reactions to macromolecular protein preparations/monoclonal antibodies, or allergies to components of the investigational drug formulation;
* 17. Active pulmonary tuberculosis;
* 18. History of immunodeficiency diseases, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
* 19. Active HBV or HCV infection or HBV/HCV co-infection;
* 20. Pregnant or lactating women;
* 21. Subjects with a known history of psychiatric drug abuse, substance abuse, or alcoholism; patients who have ceased alcohol consumption may be enrolled;
* 22. The investigator considers the subject unsuitable for participation in this clinical study due to any clinical or laboratory abnormalities or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-06-18 (Estimated); Study Completion 2028-06-19 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) is the proportion of subjects with the best overall response being CR or PR (assessed by investigator per RECIST v1.1)

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by investigator per RECIST v1.1.
ORR | Up to 24 weeks
  ORR is the proportion of subjects with the best overall response being CR or PR (assessed by IRRC per RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC per RECIST v1.1.
OS | From randomization to death from any cause (up to approximately 18 months)
  Overall Survival
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until 90 days after last dose, assessed up to 18 months
  Incidence and severity of AE determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China